CLINICAL TRIAL: NCT05212506
Title: Association of Seminal Plasma SARS-Cov19 IgG Level With Semen Parameters and Embryological Characteristics in Vaccinated Normozoospermic Men
Brief Title: Correlation Analysis of Covid-19 IgG Antibody Level in Seminal Plasma and Semen Index
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Shanghai First Maternity and Infant Hospital (Other)
Responsible Party: Principal Investigator, chen zhi qin, doctor, Shanghai First Maternity and Infant Hospital
Other Study IDs: chen008
Record Dates: First submitted 2022-01-27; First posted 2022-01-28 (Actual); Last update posted 2022-01-28 (Actual); Status verified 2022-01

CONDITIONS: Covid-19; IgG Antibody; Semen Index
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- vaccinated and unvaccinated
  Interventions: Biological: vaccinated and unvaccinated

INTERVENTIONS:
Biological: vaccinated and unvaccinated — the vaccinated :Male patients who received more than 2 injections of the covid-19 vaccine;the unvaccinated :Male patients who did not receive the covid-19 vaccine

SUMMARY:
Since December 2019, more and more cases of unexplained pneumonia appeared after exposure to the South China Seafood Market in Wuhan City, Hubei Province. Later, the disease were confirmed to be acute respiratory infectious diseases caused by the 2019 new coronavirus infection.

Even though we have had great victories in the war against this pandemic, there is still a very large number of deaths early on. As research progresses, vaccines for this infectious disease are already being developed. There are currently two vaccines in widespread use worldwide: mRNA vaccines and inactivated vaccines. In China, inactivated vaccines are more commonly used. At present, some studies believe that mRNA vaccine does not affect the pregnancy rate and abortion rate of women, but the study sample size is small, and the conclusions are limited. The effects of inactivated vaccines on fertility are still in the blank. We now hope to conduct prospective studies, mainly to study the effect of inactivated vaccine injection on male semen, and whether it has an effect on the quality of embryos in IVF patients

ELIGIBILITY:
Inclusion Criteria:

1. The man's semen quality is normal,
2. The couple meets the indications for IVF,
3. injected with the covid-19 vaccine

Exclusion Criteria:

1. In vitro fertilization due to male factors
2. Azoospermia
3. The quality of the man's semen is abnormal
4. unvacced

Ages: 22 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The man's semen quality is normal and has been injected covid-19 vaccine
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-01 (Estimated); Primary Completion 2022-03-31 (Estimated); Study Completion 2022-05 (Estimated)

PRIMARY OUTCOMES:
semen index | 2022.01-2022.03
  the semen index of the participants

SECONDARY OUTCOMES:
Fertilization rate | 2022.01-2022.04
  The percentage of eggs fertilized
embryo quality | 2022.02-2022.05
  Grading of formed embryos
clinical pregnant rate | 2022.03-2022.05
  after the embryo transplantation, calculate the pregnancy rate

CONTACTS AND LOCATIONS:
Overall Officials: zhiqin chen1, Study Director — covid-19 vaccine
Locations (1):
- Shanghai First Maternity and Infant Health Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: Undecided